CLINICAL TRIAL: NCT06946472
Title: Investigating the Impact of Metabolic Syndrome on Pain, Muscle Strength, Kinesthesia, and Functionality in Rotator Cuff Injury Rehabilitation
Brief Title: Impact of Metabolic Syndrome on Rehabilitation Outcomes in Rotator Cuff Injury
Acronym: RMY-METS
Status: Active, not recruiting | Type: Observational
Sponsor: Elif Dilara Durmaz (Other)
Responsible Party: Sponsor-Investigator, Elif Dilara Durmaz, Principal Investigator, Istinye University
Organization: Istinye University (Other)
Other Study IDs: MetS-2025-001
Record Dates: First submitted 2025-04-11; First posted 2025-04-27 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Rotator Cuff Injury (RCI); Metabolic Syndrome (MetS)
MeSH Terms: conditions — Rotator Cuff Injuries; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RCI with MetS: Participants with rotator cuff injury and diagnosed metabolic syndrome.
- RCI without MetS: Participants with rotator cuff injury but without metabolic syndrome.

SUMMARY:
This prospective comparative study aims to investigate the effect of Metabolic Syndrome (MetS) on the outcomes of a standardized rehabilitation program in patients with Rotator Cuff Injuries (RCI). Patients diagnosed with RCI will be divided into two groups based on the presence or absence of MetS, determined by NCEP-ATP III criteria. Both groups will receive the same 4-week physiotherapy protocol including hot pack, TENS, ultrasound, and therapeutic exercises. Pain intensity, pain threshold, muscle strength, kinesthesia, and shoulder functionality will be evaluated before and after treatment. The study hypothesizes that the presence of MetS negatively affects rehabilitation outcomes in patients with RCI by altering inflammation and tissue healing processes.

DETAILED DESCRIPTION:
This study aims to investigate the differences in shoulder function and rotator cuff tear outcomes between individuals with and without Metabolic Syndrome (MetS). Participants will be divided into two groups: the MetS group, which meets at least three of the NCEP-ATP III criteria for Metabolic Syndrome, and the non-MetS group, which does not have MetS.

Both groups will undergo an initial assessment, focusing on shoulder function, rotator cuff tear status, and associated factors such as age, gender, and general health conditions. The study will explore how MetS may impact the recovery and function of the shoulder in individuals with rotator cuff tears, aiming to provide insights into potential treatment and rehabilitation strategies for this population.

Data will be collected at a single time point (cross-sectional study) to evaluate baseline conditions and differences between the two groups. Statistical analyses will be performed to compare outcomes and explore potential correlations with MetS criteria.

ELIGIBILITY:
* Inclusion Criteria for the Non-MetS Group:

  * Aged between 18-65 years
  * Willing to participate in the study
  * Unilateral Rotator Cuff Tear (RMY)
* Inclusion Criteria for the MetS Group:

In addition to the above criteria, meeting at least three of the NCEP-ATP III consensus criteria for Metabolic Syndrome Stable metabolic syndrome (e.g., no significant medical changes in the last 3 months)

- Exclusion Criteria for All Participants:

* Inability to cooperate with the tests or presence of mental health issues
* Presence of cervical radiculopathy symptoms
* Presence of other orthopedic pathologies in the same shoulder (e.g., fracture, prosthesis, avascular necrosis, advanced shoulder osteoarthritis, frozen shoulder, severe scapular dyskinesia, neurological diseases, etc.)
* Presence of function-limiting neurological, vascular, or cardiac issues
* Local steroid injection to the shoulder within the last 3 months
* Receipt of physiotherapy or rehabilitation within the last 3 months
* Systemic rheumatic or inflammatory diseases
* Surgical history due to chronic rotator cuff tear
* Diagnosis of glenohumeral joint or acromioclavicular joint arthritis
* Severe scapular dysfunction or significant postural abnormalities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include individuals aged 18-65, divided into two groups:
  Non-MetS Group: Individuals with unilateral rotator cuff tear (RMY) and no Metabolic Syndrome (MetS).
  MetS Group: Individuals with unilateral RMY and MetS, defined by meeting at least three of the NCEP-ATP III criteria, with stable metabolic syndrome (no major medical changes in the last 3 months).
  Exclusion Criteria: Participants will be excluded if they have:
  Inability to cooperate or mental health issues. Cervical radiculopathy or other shoulder pathologies (e.g., fractures, arthritis).
  Recent steroid injections, physiotherapy, or surgery (within 3 months). Neurological, vascular, or cardiac disorders. Systemic inflammatory diseases or significant postural issues.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2026-03-05 (Estimated)

PRIMARY OUTCOMES:
Change in Shoulder Pain Severity (Visual Analog Scale - VAS) | Baseline and post-treatment (approximately 4 weeks)
  Pain severity will be assessed in individuals with Myofascial Pain Syndrome (MPS) affecting the shoulder using the Visual Analog Scale (VAS). The VAS is a 10 cm horizontal line where 0 indicates "no pain" and 10 indicates "worst imaginable pain." Participants will be asked to rate their pain both at rest and during common daily activities (e.g., lifting the arm, brushing hair, dressing, reaching).
  Measurements will be conducted twice: once before the treatment (baseline) and once after the intervention period to evaluate changes in pain intensity.
Change in Pain Threshold (Algometer) | Baseline and post-treatment (approximately 4 weeks)
  Pain threshold will be assessed using an algometer. The device measures the point at which pressure induces discomfort or pain. The algometer will be applied to the deltoid muscle of the affected shoulder. Participants will be asked to report when they first feel discomfort or pain, and this point will be recorded as their pain threshold. The measurement will be repeated three times for each participant, with a 30-second rest period between measurements. The average of the three measurements will be used for analysis.
  This will be measured before and after the treatment to observe any changes in pain threshold.
  Measure Type:
  Pain Threshold
  Unit of Measure:
  Pressure (in kilopascals, kPa)

SECONDARY OUTCOMES:
Change in Muscle Strength (Digital Hand Dynamometer) | Baseline and post-treatment (approximately 4 weeks)
  Muscle strength will be measured using a digital hand dynamometer to assess the strength of the shoulder's flexors, abductors, and internal/external rotators. Measurements will be performed bilaterally for comparison. The strength will be measured according to standard protocols, with patients performing the maximal force exertion during the testing.
  Each muscle group will be tested three times for accuracy, and the average of the three measurements will be used for analysis. The dynamometer will measure the maximum force exerted by the patient, and if the patient is unable to tolerate pain during the measurement, the assessment will be terminated.
  This will be measured before and after the treatment to evaluate changes in muscle strength.
  Measure Type:
  Muscle Strength (Maximum Force)
  Unit of Measure:
  Kilograms (kg) or Newtons (N)
Change in Kinesthetic Awareness (Joint Position Sense - JPS) | Baseline and post-treatment (approximately 4 weeks)
  Kinesthetic awareness (joint position sense) will be measured for the shoulder in terms of flexion and abduction. Using a digital inclinometer, the participant's ability to accurately replicate joint positions (90° flexion and 90° abduction) will be tested. The participant will close their eyes and be asked to reproduce the position of the shoulder three times for each movement. The difference between the target and the achieved angle will be recorded. The average deviation from the target angle will be used for analysis.
  This will be measured before and after the treatment to assess improvements in proprioceptive abilities.
  Measure Type:
  Joint Position Sense (JPS)
  Unit of Measure:
  Degrees (°)
Change in Shoulder Function (Quick Disabilities of the Arm, Shoulder, and Hand - Quick DASH) | Baseline and post-treatment (approximately 4 weeks)
  Shoulder function will be assessed using the Quick Disabilities of the Arm, Shoulder, and Hand (Quick DASH) questionnaire. This version of the DASH scale consists of 11 questions about the patient's ability to perform activities of daily living, specifically related to the arm and shoulder. The answers are rated from 1 (no difficulty) to 5 (unable to do). The total score is calculated by averaging the responses, subtracting 1, and multiplying by 25. A higher score indicates greater disability.
  This will be measured before and after the treatment to assess improvements in functional ability.
  Measure Type:
  Shoulder Function
  Unit of Measure:
  Score (0 to 100 scale)

CONTACTS AND LOCATIONS:
Locations (1):
- Name: Karamanoğlu Mehmetbey University Faculty of Medicine, Yunus Emre Mah. Dr. Aziz Tarhan Cad. No:21 City: Karaman Postal Code: 70200 Country: Turkey, Karaman, Turkey (Türkiye)